CLINICAL TRIAL: NCT06209398
Title: Study on the Immunogenicity and Safety of Inactivated Enterovirus Type 71 Vaccine Combined Administration With Recombinant Hepatitis B and Group A Meningococcal Vaccine
Brief Title: Immunogenicity of the Inactivated EV71 Vaccine Combined With Hepatitis B and Group A Meningococcal Vaccine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JSEPI-005
Record Dates: First submitted 2024-01-08; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Hand, Foot and Mouth Disease
MeSH Terms: conditions — Hand, Foot and Mouth Disease | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined immunization Group (Experimental): The first dose of inactivated EV71 vaccine and the third dose of hepatitis B vaccine were combined administered on day 0, and the second dose of EV71 vaccine and Group A meningococcal polysaccharide vaccine were jointly administered on day 30.
  Interventions: Biological: Enterovirus Type 71 Vaccine, inactivated ( Human Diploid Cell ); Biological: Recombinant Hepatitis B Vaccine; Biological: Group A meningococcal polysaccharide vaccine
- Single immunization Group (Active Comparator): On the 0th and 30th day, receive two doses of inactivated EV71 vaccine respectively. On the 60th day, both hepatitis B vaccine and Group A meningococcal polysaccharide vaccine were administrated.
  Interventions: Biological: Enterovirus Type 71 Vaccine, inactivated ( Human Diploid Cell )
- hepatitis B and Group A meningococcal polysaccharide vaccine Group (Active Comparator): Administrate hepatitis B vaccine on day 0, and Group A meningococcal polysaccharide vaccine on day 30.
  Interventions: Biological: Recombinant Hepatitis B Vaccine; Biological: Group A meningococcal polysaccharide vaccine

INTERVENTIONS:
Biological: Enterovirus Type 71 Vaccine, inactivated ( Human Diploid Cell ) — Used for EV71 virus susceptible individuals aged 6 months to 5 years. Each bottle (bottle) contains 0.5ml of neutralizing antibody with a potency of no less than 3.0EU for the inactivated 71 type intestinal disease vaccine. Intramuscular injection into the deltoid muscle of the upper arm. The immunization program consists of 2 doses with 1-month interval.
  Arms: Combined immunization Group; Single immunization Group
Biological: Recombinant Hepatitis B Vaccine — Each vaccine bottle (tube) is 0.5ml, containing 10ug of HBsAg and inject into the upper deltoid muscle. The immunization program consists of three doses, administered at 0, 1, and 6 months respectively. Newborns are given the first dose within 24 hours after birth, with one dose of vaccine administered each time.
  Arms: Combined immunization Group; hepatitis B and Group A meningococcal polysaccharide vaccine Group
Biological: Group A meningococcal polysaccharide vaccine — This product is made by lyophilizing the purified polysaccharide antigen obtained from Group A meningococcus liquid culture. The vaccination targets children aged 6 months to 15 years old, and the initial immunization age starts from 6 months old. Infants and young children aged 6 to 12 months old are vaccinated with 2 doses of 30 micrograms, with an interval of 3 months. Subcutaneously inject 0.5ml into the lateral deltoid muscle of the upper arm at a dose of 30 μg of polysaccharide antigen (0.5ml).
  Arms: Combined immunization Group; hepatitis B and Group A meningococcal polysaccharide vaccine Group

SUMMARY:
The main purpose of this study is to evaluate the immunogenicity and safety of inactivated enterovirus type 71 vaccine combined with recombinant hepatitis B vaccine or Group a meningococcal polysaccharide vaccine.

DETAILED DESCRIPTION:
This study conducts a randomized, controlled design, enrolled infants over 6 months old as the participant, and setting up three parallel groups. Participants are randomly assigned to three groups. The first group is the inactivated enterovirus type 71 Vaccine (EV71 vaccine), Recombinant hepatitis B vaccine and Group A meningococcal polysaccharide vaccine combined administration group. The first dose of inactivated EV71 vaccine and Recombinant hepatitis B vaccine are combined administration on day 0, and the second dose of inactivated EV71 vaccine and Group A meningococcal polysaccharide vaccine are combined administration on day 30. The second group is the inactivated EV71 vaccine single administration group, with two doses of inactivated EV71 vaccine administered on day 0 and day 30 respectively. The third group is Recombinant hepatitis B vaccine and Group A meningococcal polysaccharide vaccine administration group, the Recombinant hepatitis B vaccine is administered on day 0, and the Group A meningococcal polysaccharide vaccine is administered on day 30. Each participant will be followed up 30 minutes, 24 hours, 48 hours, and 72 hours after each vaccination actively, and will be reported for 4-30 days to collect adverse reactions/events passively. All participants collect serum samples before administration (day 0) and second dose of administration (day 30), 30 days and 1 year after full-term administration (day 60 and 1 year). The serum samples of participants will be collected 5 years after full-term administration at the first and second group. The immunogenicity of the inactivated EV71 vaccine, Recombinant hepatitis B vaccine, and Group A meningococcal polysaccharide vaccine of three groups participants will be detected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 6-7 months with no history of vaccination within the past month and normal intelligence.
* Healthy individuals determined by researchers after inquiring about medical history and physical examination.
* The recipients are able to comply with the requirements of the research protocol and undergo immunogenicity testing.
* Individuals without contraindications.
* Underarm temperature ≤ 37 ℃.
* Obtain informed consent from the recipient's guardian and sign an informed consent form.

Exclusion Criteria:

* Individuals with any serious illness.
* Individuals who are allergic to any ingredient in the research vaccine.
* Individuals with a history of neurological symptoms or signs.
* Individuals with bleeding constitution or prolonged bleeding time.
* Individuals who have had hand, foot, and mouth disease, hepatitis B, and epidemic cerebrospinal meningitis in the past.
* Individuals who have received other vaccines or immunoglobulin injections or any investigational drugs within the past 4 weeks.
* Infected individuals who have had any acute illness or require systemic antibiotic or antiviral treatment within the past 7 days.
* Individuals who have experienced fever (axillary temperature ≥ 38 ℃) within the past 3 days.
* Participating in another researcher.
* Individuals with a history or family history of allergies, seizures, epilepsy, encephalopathy, and mental illness.
* Patients with thrombocytopenia or other coagulation disorders that may cause contraindications for intramuscular injection.
* Patients with severe chronic diseases.
* Known or suspected concurrent diseases include: respiratory system diseases, acute or chronic disease activity period, HIV infection in the mother or research subject of the child, cardiovascular disease, severe hypertension, malignant tumor treatment period, and skin disease patients.
* Endemic disease patients.
* Those who plan to leave their place of residence before the end of the study.
* Researchers believe that any situation that may affect observation and evaluation.

Ages: 6 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 510 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity of inactived Enterovirus type 71 Vaccine Combined With Hepatitis B andGroup A meningococcal polysaccharide vaccine | 1 month, 1 years and 5 years after full term immunization.
  To analyze the immunogenicity after inactived EV71 vaccine, hepatitis B vaccine, Group A meningococcal polysaccharide vaccine were adminisataed after combined use and single vaccination
Safety of Enterovirus type 71 Vaccine Combined With Hepatitis B and Group A meningococcal polysaccharide vaccine | 30 minutes, 24 hours, 48 hours, and 72 hours of active follow-up, with passive reporting for 4-30 days。
  To compare the adverse reactions of inactived EV71 vaccine, hepatitis B vaccine and Group A meningococcal polysaccharide vaccine after combined use and single vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province Centers for Disease Control and Prevention, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No